CLINICAL TRIAL: NCT04859036
Title: The Effect of Transcatheter Ventricular Septal Defect Closure on Heart Rate Variability Parameters
Status: Completed | Type: Observational
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, süleyman sunkak, Principal Investigator, Kayseri City Hospital
Other Study IDs: 2014/39
Record Dates: First submitted 2021-04-20; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Ventricular Septal Defect; Closure; Interventricular Septum; Autonomic Nervous System Imbalance
Keywords: ventricular septal defect; heart rate variability; percutaneous VSD closure
MeSH Terms: conditions — Heart Septal Defects, Ventricular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transchateter VSD closure group: VSD cases treated with transcatheter closure method.
  Interventions: Diagnostic Test: 24 hours ambulatory Holter monitoring
- Control group: Healty children
  Interventions: Diagnostic Test: 24 hours ambulatory Holter monitoring

INTERVENTIONS:
Diagnostic Test: 24 hours ambulatory Holter monitoring

SUMMARY:
In this study; we evaluated the heart rate variability parameters of pediatric patients whose VSDs were closed with the transcatheter method before and after, and compared with the control group.

DETAILED DESCRIPTION:
Heart rate variability (HRV) is a sign of cardiac autonomic nervous system. Evaluation of HRV in pediatric ventricular septal defect (VSD) cases before and after transcatheter closure will enlighten us in terms of cardiac autonomic control.

Methods: 19 VSD cases treated with transcatheter closure method and 18 healthy children were enrolled in the study. 24 hours Holter rhythm monitorization was applied to all patients before closure of VSD and to the control group. In the patient group, Holter rhythm monitorization was repeated in the third months. HRV parameters were obtained from Cardio Scan Premier 12® program. Frequency domain (Total power, VLF, LF, HF, LF/HF ratio) and time domain analysis (SDNN, SDANN, SDNNi, pNN50, rMSSD) were applied.

ELIGIBILITY:
Inclusion Criteria:

* VSD diameter <6mm
* Significant left-to-right shunt
* Left atrial and ventricular enlargement detected by echocardiography or calculation of Qp/Qs ratio above 1.5 in the catheterization laboratory (Qp/Qs>1.5)

Exclusion Criteria:

* Patients with arrhythmia after the procedure
* Young patients who may be inconsistent during Holter records

Ages: 56 Months to 136 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The patient group consists of pediatric patients who underwent transcatheter VSD closure in our institute.
  The control group consists of children who admitted to our institute with the complaint of palpitations and had a normal Holter record.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Heart rate variability parameters | 24 hours
  Time Domain analysis:
  After ectopic beats and artifacts were excluded, the following indices were calculated for time domian analysis in the whole Holter recording.
  * SDNN: Standard deviation of all filtered RR intervals
  * SDANN: Standard deviation of 5-minute averages of RR intervals
  * SDNNindex: Mean of the standard deviation of all RR intervals for all the 5-minute segments
  * rMSSD: Square root of the mean of the sum of square differences between adjacent filtered RR interval
  * PNN50: Percentage of the difference between adjacent RR intervals greater than 50 milliseconds
  Frequency domain analysis:
  We determined spectral power over three frequency.
  * Very low frequency (VLF) index (0.003-0.04 Hz)
  * Low frequency (LF) index (0.04 - 0.15 Hz)
  * High frequency (HF) index (0.15 - 0.40 Hz)
  * Total power: Variance of all NN intervals approximately <0.4 Hz

CONTACTS AND LOCATIONS:
Overall Officials: Kazım Uzum, Prof., Study Chair — TC Erciyes University
Locations (1):
- Süleyman Sunkak, Kayseri, Kocasinan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Narin N, Pamukcu O, Tuncay A, Baykan A, Sunkak S, Tasci O, Uzum K, Saltik L. Percutaneous Ventricular Septal Defect Closure in Patients Under 1 Year of Age. Pediatr Cardiol. 2018 Jun;39(5):1009-1015. doi: 10.1007/s00246-018-1852-5. Epub 2018 Mar 15. PMID 29541816
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- See also: VSD closure indications — http://pubmed.ncbi.nlm.nih.gov/29541816/
- See also: Standarts of heart rate variability parameters — http://pubmed.ncbi.nlm.nih.gov/8598068/